CLINICAL TRIAL: NCT02306707
Title: Outcomes of Endoscopic Resection of Mucosal and Submucosal Lesions in the Stomach.
Acronym: OERS
Status: Completed | Type: Observational
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Other Study IDs: HREC2014/5/4.1 (3970)
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Adenoma, Villous
MeSH Terms: conditions — Adenoma, Villous | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Endoscopic Mucosal Resection: Patients who are referred for Endoscopic Mucosal Resection of Stomach Lesions will be included in this cohort.
  Interventions: Procedure: Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Endoscopic Mucosal Resection

SUMMARY:
A patient referred to have a lesion in the stomach removed. The aims of this study are to collect information on the technique of endoscopic removal of such lesions. By collecting information on a large number of patients undergoing this procedure the investigators can determine the best ways of diagnosing and removing these lesions safely and effectively.

ELIGIBILITY:
Inclusion Criteria:

* Stomach lesion > 10mm
* Lesion limited to the mucosal and/or submucosal layer (T1 lesion)
* Aged 18 years or older

Exclusion Criteria:

* Lesion less than 10mm
* Stomach lesion involves the muscularis propria (T2 lesion) on other staging modalities such as endoscopic ultrasonography (EUS)
* Aged younger than 18 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have stomach adenomas which are amendable to Endoscopic Mucosal Resection
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-10; Primary Completion 2023-03 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
Observed procedural data: Number of Participants with Adverse Events as a Measure of Safety and Tolerability Outcomes | 14 days

SECONDARY OUTCOMES:
Analysis of the costs of this procedure compared to previous treatments | 14 days
  Perform cost-utility analyses comparing different treatment approaches for stomach lesions

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bourke, MBBS, Principal Investigator — Western Sydney Local Health District
Locations (1):
- Westmead Hospital Endoscopy Unit, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Wang H, Nguyen M, Gupta S, Sidhu M, Cronin O, O'Sullivan T, Whitfield A, Lee EYT, Burgess NG, Bourke MJ. Long-term outcomes after endoscopic submucosal dissection for relative indication early gastric cancer in nonsurgical candidates. Gastrointest Endosc. 2024 Oct;100(4):647-659. doi: 10.1016/j.gie.2024.03.032. Epub 2024 Apr 3. PMID 38580133
- [Derived] Tate DJ, Klein A, Sidhu M, Desomer L, Awadie H, Lee EYT, Mahajan H, McLeod D, Bourke MJ. Endoscopic submucosal dissection for suspected early gastric cancer: absolute versus expanded criteria in a large Western cohort (with video). Gastrointest Endosc. 2019 Sep;90(3):467-479.e4. doi: 10.1016/j.gie.2019.04.242. Epub 2019 May 8. PMID 31077699